CLINICAL TRIAL: NCT01136317
Title: Comparison of Antisecretory Effect of a Single Dose of Rabeprazole 20 mg and Omeprazole 20 mg in Obese Subjects
Acronym: Oberab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Pr Stanislas Bruley des Varannes, CHU de Nantes
Other Study IDs: BRD10/1-P
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Omeprazole; Rabeprazole; Lactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Omeprazole (Experimental)
  Interventions: Drug: Omeprazole
- Rabeprazole (Experimental)
  Interventions: Drug: Rabeprazole
- Placebo (Placebo Comparator)
  Interventions: Drug: Lactose

INTERVENTIONS:
Drug: Omeprazole
  Arms: Omeprazole
Drug: Rabeprazole
  Arms: Rabeprazole
Drug: Lactose
  Arms: Placebo

SUMMARY:
This study aims to determine, in obese subjects, the antisecretory effect of a single dose of placebo, rabeprazole 20 mg and omeprazole 20 mg using 24h gastric pH monitoring, in a prospective, monocentre, randomized manner. Monitorings are separated between 6 and10 days. The main outcome criteria of analysis is the percentage of time with gastric pH above 3 during 24hours.

ELIGIBILITY:
Inclusion Criteria:

* Helicobacter negative obese subject (BMI 30 to 40),
* 18 to 55 years old,
* normal hepatic biology and morphology (echography)
* Contraceptive methods in women.

Exclusion Criteria:

* Subjects with previous abdominal surgery, with diabetic or immunosuppressive treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
In order to measure antisecretory effect, the main outcome criteria of analysis will be the percentage of time with gastric pH above 3 and measured during 24hours following rabeprazole administration in comparison with omeprazole administration.

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas Bruley des Varannes, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

REFERENCES:
- [Derived] Belhocine K, Vavasseur F, Volteau C, Flet L, Touchefeu Y, Bruley des Varannes S. Controlling on-demand gastric acidity in obese subjects: a randomized, controlled trial comparing a single dose of 20 mg rabeprazole and 20 mg omeprazole. BMC Gastroenterol. 2014 Jul 15;14:128. doi: 10.1186/1471-230X-14-128. PMID 25027286